CLINICAL TRIAL: NCT06687304
Title: Benefits of Light in the Radiographic Environment
Brief Title: Light in Healthcare Environment (Ljus i sjukhusmiljö)
Acronym: LIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: AFA Insurance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024-04436-02
Record Dates: First submitted 2024-11-04; First posted 2024-11-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sleep Quality; Well-being; Melatonin; Cortisol; Energy Levels
Keywords: Light; Radiography; Light environment; Circadian rhythm; Personnel at radiology departments
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced light environment (Active Comparator)
  Interventions: Device: Light enhancement
- Non-enhanced light environment (No Intervention)

INTERVENTIONS:
Device: Light enhancement — Light recipe that mimics the varying daylight of the day
  Other Names: Lamp; Light recipe; Dynamic lighting
  Arms: Enhanced light environment

SUMMARY:
The goal of this clinical trial is to learn if light can enhance the feeling of well-being and sleep quality in Radiographers. It will also find out if there is an optimal recipe for light. The main questions it aims to answer are:

* Will alertness, energy levels, and sleep quality increase in radiographers when the lighting is differed?
* What light recipe is the most beneficial for the personnel? Researchers will compare no enhanced light environment to different enhanced light environment to see if the enhanced light is beneficial for radiographers.

Participants will:

* Will work in an enhanced light environment or a non-enhanced light environment
* Answer surveys
* Take saliva sample

DETAILED DESCRIPTION:
The aim of this study is to examine the impact of different daylight lighting conditions in the radiographer's workplace environment. Will alertness, energy levels, well-being, and sleep quality increase in the personnel at the radiology department when the lighting is differed? Which light recipe is the most beneficial for the personnel at the radiology department? Method Design: In order to ascertain the light level that yields the desired effect, an quasi-experimental study design will be employed to identify the optimal light recipe with the appropriate light intensity. A crossover design is intended for implementation. This design approach offers the advantage of having each participant serve as their own control, thereby minimizing the potential impact of inter-group differences on the results. Furthermore, it enhances statistical efficiency, even with a reduced number of study participants (Lim & In, 2021).

Context/recruitment: Recruitments of personnel from various radiology departments at Skåne University Hospital (SUS) in Lund are planned to be conducted. A total of 18 the personnel at the radiology department will be included during the darker months of the year. At 10 to 20 workstations, a floor lamp equipped with an adjusted light prescription will be installed. Participants will be assigned to conditions in which the lamp will either be activated with the specified light recipe or remain turned off. After a duration of two weeks, the conditions will be reversed for an additional two-week period. This process will be repeated using four different light recipes to evaluate their effects on the energy levels, activity, and sleep quality of the staff. The objective is to gather insights from each season that can be implemented in the subsequent winter to determine the optimal light level.

Data collection: Subjective Measurement Methods - Staff Surveys

General Survey Participants will be asked questions regarding their typical age and gender. Additionally, a modified version of the Morningness-Eveningness Questionnaire (MEQ) will be utilized to determine each individual;s chronotype (Adan & Almirall, 1991). A Swedish translation of this questionnaire has proven effective in assessing chronotype and is appropriate for use when a shorter assessment tool is needed (Danielsson et al., 2019).

Karolinska Sleepiness Scale (KSS) To assess the level of alertness and energy among study participants, the KSS will be utilized. This scale employs a 9-point Likert format to evaluate perceived fatigue and energy levels (Åkerstedt & Gillberg, 1990). The KSS has been utilized in various research studies to examine the impact of lighting conditions on perceived alertness.

Patient-Reported Outcomes Information System Short Form Sleep Disturbance 8a(PROMIS) The Patient-Reported Outcomes Measurement Information System (PROMIS) is an assessment tool designed to measure self-reported sleep disturbances, including sleep quality, difficulty falling asleep, and staying asleep. It consists of 8 items rated by patients to evaluate the frequency and severity of sleep issues, supporting clinical insights into sleep-related health impacts.

Furthermore, participants & well-being will be quantified utilizing the WHO-5 Well-Being Index.

Objective Measurement Methods: Sleep Data via Activity Bands - Actiwatch

The employment of activity monitors allows for the objective measurement of sleep. The actigraphy device is worn on the non-dominant wrist and is non-invasive (Weiss et al., 2010). It continuously tracks the participant's movements and records sleep parameters including duration and quality. These measurements can subsequently be analyzed (Ancoli-Israel et al., 2015). Due to the impracticality of wearing these wristbands during working hours, participants will attach them to their clothing at work and wear them on their wrist after work hours.

Additionally, saliva samples will be collected to measure cortisol and melatonin levels in the study participants. Cortisol secretion is stimulated by dawn light or, in winter, often by office lighting. This secretion level provides an objective parameter for assessing activation. Conversely, melatonin secretion is suppressed by the light of dawn, and the extent of this inhibition serves as an indicator of the lights effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Radiographer

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) | Measurements will be taken three times daily over a period of 16 to 20 weeks, depending on the start date of the inclusion phase, for each period.
  To assess the subjective level of sleepiness at a particular time during the day
WHO-5 Well-Being Index | Measurements will be taken at the start and then second Friday in each two-week period over the 16 to 20 weeks (depending on when the inclusion phase can begin) during which inclusion occurs for each season.
  To assess the level of well-being, the WHO-5 Well-Being Index is used. It's a brief, self-reported measure of current mental well-being, consisting of five questions that assess positive mood, vitality, and general interest over the past two weeks.
PROMIS | Measurements will be taken at the start and then every Friday in each two-week period over the 16 to 20 weeks (depending on when the inclusion phase can begin) during which inclusion occurs for each season.
  Patient-Reported Outcomes Measurement Information System (PROMIS) is a standardized, self-reported questionnaire designed to measure an individual's perception of their sleep quality, specifically addressing issues like difficulty falling asleep, staying asleep, and feelings of restlessness. It consists of 8 items that gauge the severity of sleep disturbances over the past seven days.

OTHER OUTCOMES:
Melatonin | Measurements will be taken on Mondays, Wednesdays, and Fridays each week over the 16 to 20 weeks (depending on when the inclusion phase can begin) during which inclusion takes place for each season.
  Melatonin levels will be measured through saliva samples throughout the day to assess the variations in melatonin.
Cortisol | Measurements will be taken on Mondays, Wednesdays, and Fridays each week over the 16 to 20 weeks (depending on when the inclusion phase can begin) during which inclusion takes place for each season.
  Cortisol levels will be measured through saliva samples throughout the day to assess variations in cortisol values, allowing us to observe, e.g, variations in stress responses.

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Skånes universitetssjukhus Lund, Lund, Skåne County
  - Skånes universitetssjukhus, Malmo, Skåne County
  - Lasarettet Trelleborg, Trelleborg, Skåne County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss AR, Johnson NL, Berger NA, Redline S. Validity of activity-based devices to estimate sleep. J Clin Sleep Med. 2010 Aug 15;6(4):336-42. PMID 20726281
- [Background] Ancoli-Israel S, Martin JL, Blackwell T, Buenaver L, Liu L, Meltzer LJ, Sadeh A, Spira AP, Taylor DJ. The SBSM Guide to Actigraphy Monitoring: Clinical and Research Applications. Behav Sleep Med. 2015;13 Suppl 1:S4-S38. doi: 10.1080/15402002.2015.1046356. No abstract available. PMID 26273913